CLINICAL TRIAL: NCT03051633
Title: Substance Use Prevention Campaign for American Indian Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Randall Swaim, Senior Research Scientist, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA035141 (NIH)
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Adolescent Substance Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Be Under Your Own Influence Intervention (Experimental): School-based anti-substance use communications campaign
  Interventions: Behavioral: Be Under Your Own Influence
- Control (No Intervention): Assessment only

INTERVENTIONS:
Behavioral: Be Under Your Own Influence — School based anti-drug use communications campaign
  Arms: Be Under Your Own Influence Intervention

SUMMARY:
The goal of this project is to test the effectiveness of a successful anti-drug communications campaign (Be Under your Own Influence) to lower substance use among AI 7th graders. The campaign uses messages that support youths' personal autonomy and future aspirations, and these messages are delivered to 7th graders using high school students. Our goal is to develop a turnkey package for the broader population of AI youth and schools and to develop components that can incorporate flexibility and creativity in their delivery.

DETAILED DESCRIPTION:
Substance use is a particularly dangerous risk to middle-school youth, and American Indian (AI) youth are at increased risk. We have found over the course of more than three decades that substance use among AI youth is consistently higher than that of other ethnic/racial groups.

Schools are often the site for adolescent drug prevention efforts, but results from these efforts are often modest or even disappointing. This intervention adapts an existing campaign (Be Under Your Own Influence; BUYOI) that has been found to be effective in reducing substance use and that uses campaign messages that are congruent with AI culture. The intervention will be adapted using significant contributions from tribal members, including youth, teachers, parents, elders, and other community members. This proposal includes active involvement of local advisory boards, hiring of a local AI liaison, focus groups, a youth photo voice component, and use of AI staff from our Center and from the Native American Cultural Center at our university.

The adapted anti-drug and alcohol use communications campaign will be delivered by selected high school students to 7th grade students. A distinguishing feature of the BUYOI campaign is a message that targets outcome expectations related to aspirations, autonomy, and physical harms. The campaign will use multiple channels of communication including print (e.g., posters and fliers), video and audio spots, presentations, and social media to deliver messages that are designed to alter outcome expectancies, intentions, and ultimately substance use among targeted youth.

The campaign will be delivered to two cohorts of 7th graders, with 4 longitudinal measurement occasions for each cohort. Five middle schools (and their corresponding high schools) have been recruited for the study, where three of these will be randomly assigned to the intervention condition and two to the control condition. Multilevel data analysis will test for effects of campaign exposure on autonomy, aspirations, perceived harm, and intentions to use.

Because of the heavy involvement of the school and community in the development and delivery of the intervention, we will be able to incorporate sustainability into the design of all integrated components. Ultimately, our goal is to develop a turnkey package for the broader population of reservation-based AI youth and schools and to develop components that can incorporate flexibility and creativity in their delivery. For example, a school or local group may implement the campaign in its original form or they may modify aspects to make them more pertinent to their community.

ELIGIBILITY:
Inclusion Criteria:

* Attend 7th grade in targeted schools that are on or near American Indian reservation and have received parental consent

Exclusion Criteria:

* No parental consent

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2014-04-15 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Be Under Your Own Influence Intervention | Control
Started | 342 | 186
Completed | 249 | 179
Not Completed | 93 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Be Under Your Own Influence Intervention | Control | Total
Number analyzed (Participants) | 342 | 186 | 528
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 342 | 186 | 528
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age not reported by respondent.
  Years
    number analyzed (Participants) | 248 | 164 | 412
    (all) | 12.5 (.57) | 12.5 (.65) | 12.5 (.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data was not given by the respondent.
  Participants
    number analyzed (Participants) | 339 | 186 | 525
    Female | 188 | 91 | 279
    Male | 151 | 95 | 246
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 47 | 65
  Not Hispanic or Latino | 324 | 139 | 463
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 321 | 176 | 497

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Initiation
Description: The number of students who self-reported initiated alcohol for the first time during the study period
Time Frame: 18 months
Population: BUYOI efficacy was tested in a five-year study with two cohorts of middle school students, and five middle schools recruited from the Northern Plains and Southwest regions of the United States, representing a recent sample of American Indian adolescents (grades 7th-8th, age at first assessment = 12.5 years).
Measure: Count of Participants; unit: Participants
Arm/Group | Be Under Your Own Influence Intervention | Control
Number analyzed (Participants) | 342 | 186
Participants | 160 | 109
Statistical Analysis 1: Comparison: Be Under Your Own Influence Intervention; Discrete time hazard represents the conditional probability that a student will experience first time alcohol use during a given measurement period, given that students did not use alchohol in a previous measurement period. Thus for each model, we tested the following hypothesis: Controlling for age at first-assessment, students attending BUYOI-assigned schools will have a lower risk of substance use uptake by the end of their eighth-grade year, relative to students attending control schools; Test type: Superiority — Event: Dichotimized self-reported first-time alcohol use in known participant history prior to data-collection, where substance use was not previously reported in prior measurement occasions of this four-wave longitudinal study. Episodes: Episodes represent the period of time between measurement occasions, as such, each episode represents the measured period of time between each wave of assessments. Censoring: If substance use was reported, censoring indicator indicates the risk period; p = .004, Regression, Logistic; Discrete time hazard model represents a survival analysis, with the outcome parameters reflecting a hazard ratio rather than odds; Hazard Ratio (HR) = -0.42, 95% CI 2-sided [-0.714 to -0.126]

2. Primary Outcome: Alcohol Intoxication Initiation
Description: Number of participants self-reporting first-time alcohol intoxication initiation during the study period.
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Be Under Your Own Influence Intervention | Control
Number analyzed (Participants) | 342 | 186
Participants | 90 | 62
Statistical Analysis 1: Comparison: Be Under Your Own Influence Intervention; Discrete time hazard represents the conditional probability that a student will experience first time alcohol initiation during a given measurement period, given that students did not become intoxicated in a previous measurement period. Thus, for each model, we tested the following hypothesis: controlling for age at first assessment, students attending BUYOI-assigned schools will have a lower risk of substance use uptake at the end of their eight grade year; Test type: Superiority — Event: dichotimized self-reported first-time alcohol intoxication in known participant history prior to data collection, where intoxication was not reported in prior measurement occasions. Episodes: Represent the period of time between measurement occasions, thus, each episode represents the measured period of time between each assessment wave. Censoring: Indicates the risk period during which particpants experienced intoxication uptake; p = .037, Regression, Logistic; Discrete time hazard model represents a survival analysis, with the outcome parameters reflecting a hazard ration rather than odds; Hazard Ratio, log = -0.39, 95% CI 2-sided [-0.762 to -0.018]

3. Primary Outcome: Marijuana Initiation
Description: Number of participants who self-reported first-time marijuana use initiation during the study period
Time Frame: 18 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Be Under Your Own Influence Intervention | Control
Number analyzed (Participants) | 342 | 186
Participants | 183 | 97
Statistical Analysis 1: Comparison: Be Under Your Own Influence Intervention vs Control; Discrete time hazard represents the conditional probability that a student will experience first time marijuana use during a given measurement period, given that students did not use marijuana in a previous measurement period. Thus for each model, we tested the following hypothesis: Controlling for age at first-assessment, students attending BUYOI-assigned schools will have a lower risk of marijuana use uptake by the end of their eighth-grade year, relative to students attending control schools; Test type: Superiority — Event: Dichotimized self-reported first-time marijuana use in known participant history prior to data-collection, where marijuana use was not previously reported in prior measurement occasions of this four-wave longitudinal study. Episodes: Episodes represent the period of time between measurement occasions, as such, each episode represents the measured period of time between each wave of assessments. Censoring: If marijuana use was reported, censoring indicator indicates the risk period; p = 0.228, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Hazard Ratio, log = 0.17, 95% CI 2-sided [-0.104 to 0.444]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Be Under Your Own Influence Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/342 | 0/186
Serious Adverse Events (participants affected / at risk) | 0/342 | 0/186
Other Adverse Events (participants affected / at risk) | 0/342 | 0/186

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT03051633/Prot_SAP_000.pdf